CLINICAL TRIAL: NCT05294237
Title: Injury Prevention in Danish Youth Handball - a Hybrid Effectiveness-implementation Study
Brief Title: Injury Prevention in Danish Youth Handball
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Handball Federation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDU-2021-57-(2089)
Record Dates: First submitted 2021-06-24; First posted 2022-03-24 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Adherence, Sports Injury Prevention Exercises; Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Palliative Care

STUDY DESIGN:
Masking Description: The clubs will be randomly assigned to either the control or intervention group at a 1:1 allocation ratio, using a computer-generated randomisation schedule. The randomisation will be performed by a person not else involved in the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Implementation (Intervention) (Experimental): The Happy-program will be available online on a webpage and consists of 7 warm-up components and 4 resistance training components that can be completed after handball practice.
  The warm-up program has three exercise variations for each of the seven components. The coaches may deliver the four resistance training components in the field or in the gym. The resistance training components in the field and the gym targets the same four body areas but differs in that the components in the gym are performed with equipment, while the components in the field can be performed without equipment. Each resistance training component has three levels.
  Happy ambassadors (Health professionals with a handball player or coach background) will conduct a 3-hour train-the trainer workshop in the beginning of the season and provide coaches with the opportunity for support throughout the season. At mid-season, the ambassadors will re-visit the clubs for 1,5-hour supervision and support.
  Interventions: Behavioral: Happy program; Behavioral: Support
- Unsupported implementation (control) (Active Comparator): Access to the Happy program will be available online to the coaches. No additional education or support will be provided.
  Interventions: Behavioral: Happy program

INTERVENTIONS:
Behavioral: Happy program — The Happy program consists of handball specific warm-up components and resistance training components and will be available online.
Behavioral: Support — The support consists of a coach workshop at the beginning of the season and the opportunity for additional support for the coaches throughout the season.
  Arms: Supported Implementation (Intervention)

SUMMARY:
The primary aim of this hybrid-effectiveness-implementation cluster randomised study is to investigate if a supported implementation of an injury prevention exercise program (Happy program) involving a train-the-trainer workshop and coach support during the season is superior to an unsupported implementation of the Happy program involving the availability of the program on webpages, in improving adherence (volume, frequency, duration) of the Happy program among coaches for young (11-17 years of age) Danish female and male handball players during one handball season. Secondary aims are to investigate if the supported implementation is superior to the unsupported implementation in improving behavioural outcomes among the coaches and in reducing the risk for new ankle, knee, and shoulder injuries among young (11-17 years of age) Danish female and male handball players during one handball season. Further, the investigators aim to evaluate how and why adherence and behavioural determinants towards use of the Happy program might improve (or not).

ELIGIBILITY:
Inclusion Criteria:

* playing in youth teams from the age groups under (u)13, u15, and u17
* playing in handball club with at least four teams in the desired age groups

Exclusion Criteria:

-

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female, male, non-binary, prefer not to answer, other
Enrollment: 950 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence volume at team level | Measured weekly over 7 months
  How much the Happy components have been delivered (adherence volume) will be evaluated as the number of Happy components delivered per week at team level over the full season
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week
Shoulder, knee and ankle injuries using the Oslo Sports Trauma Research Center Health problems Questionnaire (OSTRC-H2) | Measured weekly over 7 months
  The primary injury outcomes will be time to any new handball-related ankle, knee and shoulder injury defined as any tissue damage or other derangement of normal physical function due to participation in handball, resulting from rapid or repetitive transfer of kinetic energy, following a recent consensus statement from the International Olympic Committee
  Injury status will be monitored weekly during the season using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application. The questionnaire also measures exposure to handball, both training and match, during the last seven days.

SECONDARY OUTCOMES:
Adherence volume of the Happy warm-up components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the warm-up components included in the Happy program, an evaluation of how much the Happy warm-up components have been delivered at team level will be evaluated as the number of Happy warm-up components delivered per week over the full season
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week
Adherence volume of the Happy resistance training components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the resistance training components included in the Happy program, an evaluation of how much the Happy resistance training components have been delivered at team level will be evaluated as the number of Happy resistance training components completed per week over the full season
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week
Adherence volume of the Happy resistance training components at player level | Assessed weekly over 7 months
  To support the evaluation at team level, an evaluation of how much the Happy resistance training components has been completed will be evaluated at player level as the number of Happy resistance training components completed per week over the full season
  Reports of Happy resistance training components usage will be recorded electronically on a weekly basis by the player using an application.
Substantial shoulder, knee and ankle injuries using the Oslo Sports Trauma Research Center Health problems Questionnaire (OSTRC-H2) | Assessed weekly over 7 months
  Secondary injury outcomes will be time to any substantial handball related ankle, knee and shoulder injury.
  Injuries will be defined as any tissue damage or other derangement of normal physical function due to participation in handball, resulting from rapid or repetitive transfer of kinetic energy, following the 2020 consensus statement from the International Olympic Committee. Players reporting at least a moderate reduction in training volume or performance due to a health problem with the Oslo Sports Trauma Research Center Health Questionnaire and further classify the health problem as a new shoulder, knee or ankle injury is defined as an substantial injury.
  Injury status will be monitored weekly during the season using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application. The questionnaire also measures exposure to handball, both training and match, during the last seven days.
Health Action Process Approach (HAPA) Questionnaire responses | Will be assessed at baseline, mid-season (3 months after baseline) and at end season (7 months)
  A questionnaire will be used to assess between-group differences in HAPA constructs (ie: intentions, outcome expectancies, self-efficacy, action planning and coping planning) between baseline and the mid-season and the end of playing season.
Determinants of Implementation Behavior Questionnaire (DIBQ) responses | Will be assessed at baseline, mid-season (3 months after baseline) and at end season (7 months)
  To support the Health Action Process Approach (HAPA) Questionnaire responses, The Determinants of Implementation Behavior Questionnaire (DIBQ) constructs focusing on social influences will be measured at baseline, at mid-season and at the end of the season. These questions will be added to the same questionnaire assessing the HAPA constructs.

OTHER OUTCOMES:
Training volume | Assessed weekly over 7 months
  Number of training hours will be used to assess the player's exposure to handball training.
  Will be assessed weekly as a add on to the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application.
Match volume | Assessed weekly over 7 months
  Number of match hours will be used to assess the player's exposure to handball matches.
  Match volume will be assessed weekly as a add on to the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application.
Illness outcomes using the Oslo Sports Trauma Research Center Health problems Questionnaire (OSTRC-H2) | Assessed weekly over 7 months
  Illness will be defined is a complaint or disorder experienced by an athlete, not related to the injury. Illnesses include health- related problems in physical (eg, influenza), mental (eg, depression), or social well-being or removal or loss of vital elements (air, water, warmth), following the 2020 consensus statement from the International Olympic Committee.
  Illness status will be monitored weekly during the season using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application. The questionnaire also measures exposure to handball, both training and match, during the last seven days.
Injury outcomes using the Oslo Sports Trauma Research Center Health problems Questionnaire (OSTRC-H2) | Assessed weekly over 7 months
  Other injury outcomes will be all injuries.
  Injuries will be defined as any tissue damage or other derangement of normal physical function due to participation in handball, resulting from rapid or repetitive transfer of kinetic energy, following the 2020 consensus statement from the International Olympic Committee.
  Injury status will be monitored weekly during the season using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire distributed electronically to the players via an application. The questionnaire also measures exposure to handball, both training and match, during the last seven days.
Adherence duration at team level | Assessed weekly over 7 months
  How long the Happy components have been delivered (adherence duration) will be evaluated as the proportion of all possible weeks where Happy components are delivered at team level over the full season.
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week.
Adherence duration of the the Happy warm-up components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the warm-components included in the Happy program, an evaluation of for how long Happy warm-up components have been delivered at team level will be evaluated as the proportion of all possible weeks where Happy warm-up components are delivered at team level over the full season.
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week.
Adherence duration of the Happy resistance training components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the resistance training components included in the Happy program, an evaluation of for how long the Happy resistance training components have been delivered will be evaluated evaluated as the proportion of all possible weeks where Happy resistance training components are delivered at team level over the full season.
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week.
Component fidelity at team level | Assessed weekly over 7 months
  The number of each Happy component completed of total number of each recommended over the season.
Adherence duration of the Happy resistance training components at player level | Assessed weekly over 7 months
  To support the evaluation at team level, an evaluation of for how long the Happy resistance training components has been completed will be evaluated at player level as the proportion of all possible weeks where Happy resistance training components are completed at player level over the full season.
  Reports of Happy resistance training components usage will be recorded electronically on a weekly basis by the player using an application.
Adherence frequency at team level | Assessed weekly over 7 months
  How frequently the Happy components have been delivered (adherence frequency) will be evaluated as the average times per week Happy components were delivered at team level over the full season
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week
Adherence frequency of the Happy warm-up components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the warm-components included in the Happy program, an evaluation of how frequently the Happy warm-up components have been delivered will be evaluated as the average times per week Happy warm-up components were delivered at team level over the full season.
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week.
Adherence frequency of the Happy resistance training components at team level | Assessed weekly over 7 months
  To gain a detailed understanding of the adherence to the resistance training components included in the Happy program, an evaluation of how frequently the Happy resistance training components have been delivered will be evaluated as the average times per week Happy resistance training components were delivered at team level over the full season.
  Reports of Happy program usage will be recorded electronically on a weekly basis by the head coach of each team using a web application. A full warm-up session includes 7 components. A full resistance exercise training includes 4 components. The coaches are encouraged to perform all Happy program components with their players twice a week.
Adherence frequency of the Happy resistance training components at player level | Assessed weekly over 7 months
  To support the evaluation at team level, an evaluation of how frequently the Happy resistance training components has been completed will be evaluated at player level as the average times per week Happy resistance training components were completed at player level over the full season.
  Reports of Happy resistance training components usage will be recorded electronically on a weekly basis by the player using an application.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Møller, PhD, Principal Investigator — University of Southern Denmark, Department of Sports Science and Biomechanics
Locations (1):
- University of Southern Denmark, Odense, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller M, Nygaard Andersen L, Moller S, Kongsted A, Juhl CB, Roos EM. Health And Performance Promotion in Youth (HAPPY) hybrid effectiveness-implementation cluster randomised trial: comparison of two strategies to implement an injury prevention exercise programme in Danish youth handball. Br J Sports Med. 2024 Oct 22;58(20):1205-1214. doi: 10.1136/bjsports-2023-107880. PMID 39209524